CLINICAL TRIAL: NCT05487495
Title: First-in-Human (FIH), Open-Label, Non-Randomized, Single-Arm Phase 1 Study to Evaluate the Safety and Tolerability of Donor-Derived CD5 CAR T (CT125B) Cells ForRelapsed or Refractory T-Cell Acute Lymphoblastic Leukemia/Lymphoma
Brief Title: Donor-Derived CD5 CAR T (CT125B) Cells for Relapsed or Refractory T- Cell Acute Lymphoblastic Leukemia/Lymphoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: ethic commitee decisiong
Sponsor: Beijing Boren Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRYY-IIT-LCYJ-2022-026
Record Dates: First submitted 2022-08-01; First posted 2022-08-04 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2022-08

CONDITIONS: T-Cell Acute Lymphoblastic Leukemia/Lymphoma
Keywords: CAR-T; Leukemia; acute lymphoblastic leukemia/lymphoma
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma; Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CD5 CAR T (CT125B) (Experimental): All patients who receive CD5 CAR T (CT125B) cell infusion.
  Interventions: Biological: CD5 CAR T (CT125B)

INTERVENTIONS:
Biological: CD5 CAR T (CT125B) — Subjects will be pretreated with chemotherapy prior to infusion of CAR T cells: After the collection of PBMC and about 5 days before infusion, lymphodepletion (fludarabine at 30 mg/m^2/day and cyclophosphamide at 250 mg/m^2/day; for prior-SCT donor-derived CAR T-cell infusion) or intensified lymphodepletion (fludarabine at 30 mg/m^2/day and cyclophosphamide at 30 mg/kg/day; for new donor-derived CAR T-cell infusion) will be administrated for 3 days.

SUMMARY:
This is a FIH, single center, open label, non-randomized, single-arm, Phase I clinical trial to evaluate the safety and tolerability of CD5 CAR T (CT125B) cells in subjects with relapsed or refractory T-cell acute lymphoblastic leukemia/lymphoma. 9-18 subjects will be enrolled. After the collection of PBMC and about 5 days before infusion, lymphodepletion (fludarabine at 30 mg/m^2/day and cyclophosphamide at 250 mg/m^2/day; for prior-SCT donor-derived CAR T-cell infusion) or intensified lymphodepletion (fludarabine at 30 mg/m^2/day and cyclophosphamide at 30 mg/kg/day; for new donor-derived CAR T-cell infusion) will be administrated for 3 days.

Then this study will be using BOIN1/2 approach from starting dose 1: 1×10^6 (±20%) to dose 2: 2×10^6 (±20%). If the manufactured cells were not sufficient to meet the preassigned standard dose criteria, patients are given infusion at a low dose of 5×10^5 (±20%) /kg.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Candidates with relapsed or refractory CD5+ T cell acute lymphoblastic leukemia/lymphoma, who have progressed after treatment with all standard therapies or been intolerant of standard care, have limited prognosis with currently available therapies and had no available curative treatment options (such as SCT or chemotherapy)
2. Male or female, aged 1-70 years
3. No serious allergic constitution
4. Eastern Cooperative Oncology Group (ECOG) performance status (Oken et al., 1982) score 0 to 2
5. Have life expectancy of at least 60 days based on investigator's judgement
6. CD5 positive on blasts in bone marrow or CSF by flow cytometry, or CD5 positive on tumor tissues by immunohistochemistry; (CD5 positive criteria: Flow cytometry: Positive: > 80% of tumor cells expressed CD5 and the mean fluorescence intensity (MFI) of CD5 is the same as that in normal T cells; Dim: > 80% of tumor cells expressed CD5, but the MFI of CD5 is lower than that in normal T cells as least as 1 log; Partial positive: 20-80% of tumor cells expressed CD5 and the MFI of CD5 is the same as that in normal T cells. Tumor tissue immunohistochemistry: Positive > 30% tumor cells expressed CD5)
7. Provide a signed informed consent before any screening procedure. Patients who voluntarily participate in the study should have the ability to understand and sign the informed consent form (ICF) and be willing to follow the visit schedule and relevant study procedure, as specified in the protocol. Candidates aged 19-70 years old need to be sufficiently conscious and able to sign the treatment consent form and voluntary consent form. Candidates of 8-18 years old need to be sufficiently conscious and able to sign the treatment consent form and voluntary consent form, besides, their legal guardian or patient advocate also need to sign the treatment consent form and voluntary consent form. Children candidates of 1-7 years old can be recruited after the legal guardian or patient advocate need to sign the treatment consent form and voluntary consent form.
8. Have suitable and available allogeneic hematopoietic stem cell transplantation donor, and is willing to proceed to SCT if achieve CR.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Intracranial hypertension or disorder of consciousness
2. Symptomatic heart failure or severe arrhythmia
3. Symptoms of severe respiratory failure
4. Complicated with other types of malignant tumors
5. Diffuse intravascular coagulation
6. Serum creatinine and / or blood urea nitrogen ≥ 1.5 times of the normal value
7. Suffering from septicemia or other uncontrollable infections
8. Patients with uncontrollable diabetes
9. Severe mental disorders
10. Obvious and active intracranial lesions were detected by cranial magnetic resonance imaging (MRI)
11. Have received organ transplantation (excluding bone marrow transplant)
12. Reproductive-aged female patients with positive blood HCG test
13. Screened to be positive of infection of hepatitis (including hepatitis B and C), AIDS or syphilis
14. Post-CAR SCT is not feasible in patients
15. No donor is applicable for peripheral blood mononuclear cell (PBMC) collection or no frozen donor's PBMC is available for manufacturing CAR T cells.
16. Patients unable to discontinue nucleoside antiviral drugs that have a similar mechanism to ganciclovir

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence and type of dose-limiting toxicity (DLT) | 21 days post intravenous injection
  DLT assessment according to the clinical study protocol.
Incidence and severity of adverse events (AE) | 30 days post intravenous injection
  Incidence and severity of adverse events as assessed by NCI-CTCAE 5.0.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 30 days post infusion
  Objective response rate (ORR) according to NCCN.
Counts and persistence of CAR T cells | 30 days post infusion
  Blood samples for determination of persistence/counts of infused CAR T cells will be analysed.
Incidence and grade of severe adverse events (SAEs) | 2 years post infusion
  Incidence and severity of severe adverse events as assessed by NCI-CTCAE 5.0.
Best overall response (BOR) rate | 3 months post infusion
  Best overall response (BOR) rate according to NCCN.
The counts of CART cells after using CAR T suicidal switch drugs . | 7 days post administration of ganciclovir
  The counts of CART cells change when CAR T suicidal switch drugs ( ganciclovir ) are used for 3 days and 7 days respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Pan, MD/PhD, Principal Investigator — Beijing Gaobo Boren Hospital
Locations (1):
- Beijing Gaobo Boren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No